CLINICAL TRIAL: NCT06621771
Title: A Piano Training Program to Improve Manual Dexterity and Upper Extremity Function in Subacute Stroke Survivors
Brief Title: Playing Piano to Improve Hand Function Early After Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University (Other)
Collaborators: Jewish Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, Anouk Lamontagne, Associate Professor, McGill University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MP-50-2024-2096
Record Dates: First submitted 2024-09-25; First posted 2024-10-01 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Stroke
Keywords: Music therapy; Rehabilitation; Intervention; Upper extremity; dexterity
MeSH Terms: conditions — Stroke | interventions — Occupational Therapy

STUDY DESIGN:
Intervention Model Description: Experimental study involving a repeated-measure designed of two groups of participants with stroke, i.e., those receiving piano training sessions and those receiving additional conventional occupational therapy sessions.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Piano group (Experimental): Participants will engage in a step-by-step musical training consisting of two supervised, individual 45-min sessions per week for 6 consecutive weeks, for a total of 12 sessions. They will also be asked to practice 2x/week for 15 minutes and they will report on their practice duration and content in a logbook after each practice session.
  Interventions: Other: Music intervention
- Conventional group (Active Comparator): Participants will engage in two supervised and individual 45-min session per week for 6 consecutive week, consisting in usual occupational therapy treatment. They will be asked to practice 2x/week for 15 minutes and they will report on their practice duration and content in a logbook after each practice session.
  Interventions: Other: Occupational Therapy

INTERVENTIONS:
Other: Music intervention — Participants will engage in a step-by-step piano training consisting in playing piano pieces designed to involve all 5 digits of the paretic hand and increasing in complexity. They will be using a Musical Instrument Digital Interface (MIDI) piano program called Synthesia to display musical pieces on a computer screen that is adapted for people with no music reading abilities and will be playing on a touch sensitive piano keyboard. The supervised session will also be complemented with a unsupervised home program consisting of piano sequence exercises comprising short excerpts of the same musical pieces practiced during the supervised sessions and they will receive a roll-up flexible piano
  Arms: Piano group
Other: Occupational Therapy — Participants will receive conventional occupational therapy treatment (e.g., mobility, ADL, IALD, information session), excluding treatments focusing specifically on arm and hand motor recovery.The supervised session will also be complemented with an unsupervised home program consisting of assignments related to occupational therapy exercises and/or IALD/ADLs.
  Arms: Conventional group

SUMMARY:
The goal of this clinical trial is to study the feasibility of a 6-week piano playing training intervention in a subacute stroke population. More specifically, the investigators aim to (1) implement and test the feasibility of the intervention in the subacute stroke rehabilitation program; and (2) explore the acceptability of the supervised training sessions and home practice sessions. Researchers will also (3) estimate and contrast the effects of the piano training intervention as compared to conventional therapy on manual dexterity, coordination, functional use of the upper extremity, attention and mood.

Therapy specifically provided as part of this project will be delivered above and beyond usual therapy time in both intervention groups. Participants of the piano group will:

* Engage in a step-by-step musical training consisting of two supervised, individual 45-min sessions per week for 6 consecutive weeks, for a total of 12 sessions.
* The supervised session will also be complemented with a biweekly home program (15 minutes) consisting of piano exercises.

Participants in the conventional group will:

* Engage in two individual 45-min sessions per week for 6 consecutive weeks consisting in conventional occupational therapy treatment.
* They will also receive a biweekly home program consisting in occupational therapy exercises (15 minutes).

DETAILED DESCRIPTION:
Piano Training: Musical pieces are designed to involve all 5 digits of the paretic hand. Whether played with the right or left hand, they involve the same number of finger repetitions as well as similar finger sequences and melodic patterns. A Musical Instrument Digital Interface (MIDI) piano program called Synthesia will be used to display musical pieces on a computer screen that is adapted for people with no music reading abilities. Participants will be cued to press a sequence of key presses required to produce a melody by a visual display showing a blue dot falling from the upper part of the screen down to indicate the correct key on a virtual keyboard. After each cue, the program will pause until the participant pressed the correct key before moving on. During the supervised training sessions, participants will play on a touch sensitive piano keyboard. A computer will record the responses from the piano keyboard and provided a final score indicating the number of errors and total duration for each musical piece. A professional therapist will be present during these supervised sessions and will provide verbal feedback on the quality of movement and discouraged compensatory strategies. Nine musical pieces will be introduced to the participants in an order of increasing difficulty: level 1 involving movements of consecutive fingers (e.g.,1-2-3-4-5); level 2 involving third, fourth, and fifth intervals or movements of non-consecutive fingers (e.g., 1-3-5-1-4); and level 3 involving chords, that is 2 fingers played at the same time. Within each level, 3 musical pieces involving an increasing number of key presses and changes in melodic direction will be introduced. The speed of execution or tempo will also increase within each musical piece.

Conventional Intervention: Conventional sessions will consist of usual occupational therapy treatment (e.g., mobility, ADL, IALD, information session), excluding treatments focusing specifically on arm and hand motor recovery. The nature therapy provided as part of the conventional intervention will be carefully documents in the chart.

Home Practice: All participants in the piano group will receive an unsupervised home program consisting of piano sequence exercises comprising short excerpts of the same musical pieces practiced during the supervised sessions and they will receive a roll-up flexible piano. Participants in the conventional group will receive assignments related to occupational therapy exercises and/or IALD/ADLs. All participants will report on their practice duration and content in a logbook after each practice session.

ELIGIBILITY:
Inclusion Criteria:

* Have normal/corrected visual and auditory acuity
* Present a first-ever supratentorial unilateral stroke (1-24 weeks post-stroke)
* Present some capacity of dissociation of arm and finger movements, as reflected by scores of 3 to 6 on the arm and hand components of the Chedoke McMaster Stroke Assessment
* Have the capacity to follow simple instructions
* Have no professional piano experience (only for the piano group)

Exclusion Criteria:

* Presence of visual field defect, hemineglect as well as dementia or moderate-to-severe cognitive deficits (score less than 18 on the Montreal Cognitive Assessment).

Ages: 40 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-10-15 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Feasibility: Characteristics of stroke participants | Pre-intervention (week0)
  Collected via chart review (e.g. CPA vs. outpatient program, age, sex/gender, stroke characteristics, upper extremity function level, cognitive function)
Feasibility: Number of eligible vs. referred participants | Post-intervention (week6)
  Assessed using the number of participants referred to the study in comparison to the list of admitted patients in the targeted stroke programs.
Feasibility: adherence to intervention - number of completed sessions | Post-intervention (week6)
  Training logbook filled by researchers/clinicians (supervised sessions) and subjects (unsupervised sessions).
Feasibility: adherence to intervention - number of piano pieces completed (piano group) vs occupational therapy exercises completed (conventional group) | Post-intervention (week6)
  Training logbook filled by researchers/clinicians (supervised sessions) and subjects (unsupervised sessions).
Feasibility: adherence to intervention - number of home practice sessions | Post-intervention (week6)
  Training logbook filled by researchers/clinicians (supervised sessions) and subjects (unsupervised sessions).
Feasibility: adherence to intervention - time of home practice sessions | Post-intervention (week6)
  Training logbook filled by researchers/clinicians (supervised sessions) and subjects (unsupervised sessions).
Feasibility: presence of adverse or undesirable effects during the intervention | Post-Intervention (week6)
  Collected with open-ended questions.
Acceptability of the intervention | Post-intervention (week6)
  Participant's comments and observations collected using the Theoretical Framework of Acceptability (TFA) Questionnaire, which considers different dimensions such as affective attitude, perceived effectiveness, ethicality and opportunity cost. It comprises 8 items rated from 1 to 5. Minimum value is 8 and maximum value is 40. A higher score is associated with better outcomes.
Acceptability: Overall experience | Post-intervention (week6)
  Investigated through open-ended questions

SECONDARY OUTCOMES:
Change from Baseline in the Box and Block test at Post-intervention | Post-intervention (week6) and Follow-up (week12)
  Assess gross manual dexterity
Change from Baseline in the Nine Hole Peg Test (NHPT) at Post-intervention | Post-intervention (week6) and Follow-up (week12)
  Assesses fine manual dexterity
Change from Baseline in the Finger to Nose test at Post-intervention | Post-Intervention (week6) and Follow-up (week12)
  Assesses arm movement coordination.
Change from Baseline in the Finger Tapping test at Post-intervention | Post-intervention (week6) and Follow-up (week12)
  Assesses finger movement coordination.
Change from Baseline in the 6-items Jebsen Hand Function test at Post-intervention | Post-intervention (week6) and Follow-up (week12)
  Assesses functional use of the upper extremity.
Change from Baseline in the Digit Span Test - Forward at Post-intervention | Post-intervention (week6) and Follow-up (week12)
  A subtest of the Wechsler Adult Intelligence Scale-Fourth Edition (WAIS-IV) that assesses attention, more specifically auditory recall and working memory. Score is calculates as the longest number of forward sequential digits that can accurately be remembered. The maximum score is 16. A higher score is associated with better outcomes.
Change from Baseline in the Digit Span Test - Backward at Post-intervention | Post-intervention (week6) and Follow-up (week12)
  A subtest of the Wechsler Adult Intelligence Scale-Fourth Edition (WAIS-IV) that assesses attention, more specifically auditory recall and working memory. Score is calculates as the longest number of backward sequential digits that can accurately be remembered. The maximum score is 16. A higher score is associated with better outcomes.
Change from Baseline in the Hospital Anxiety and Depression Scale at Post-intervention | Post-intervention (week6) and Follow-up (week12)
  A self-administered test assessing mood, more specifically screening for depression and anxiety. It comprises 14 items rated from 0 to 3. Seven questions relate to anxiety and seven to depression, giving two scores (maximum score for each = 21). A higher score is associated with worse outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Anouk Lamontagne, PhD, Principal Investigator — McGill University
Locations (1):
- Jewish Rehabilitation Hospital, Laval, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available.
Time Frame: Data will be available within 6 months after study completion
Access Criteria: Data will be made available to other researchers via an institutional data repository that will allow adhering to FAIR principles.

DOCUMENTS (1):
  • Informed Consent Form (2024-10-01): https://cdn.clinicaltrials.gov/large-docs/71/NCT06621771/ICF_001.pdf